CLINICAL TRIAL: NCT02526186
Title: Battlefield Auricular Acupuncture for Control of Post-partum Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FWH20150072H
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Results first posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-02

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard of Care (No Intervention): Standard of Care only
- Battlefield Auricular Acupuncture (Experimental): Standard of Care plus Battlefield Auricular Acupuncture
  Interventions: Device: Battlefield Auricular Acupuncture

INTERVENTIONS:
Device: Battlefield Auricular Acupuncture
  Arms: Battlefield Auricular Acupuncture

SUMMARY:
We will conduct a randomized controlled trial to determine whether the addition of battlefield auricular acupuncture to standard of care is effective for control of postpartum pain for mothers in the immediate post-partum period. Post-partum patients (DoD beneficiaries) 18 years or older, regardless of gravida/parity, who plan to have a childbirth in a hospital setting will be offered the opportunity to participate in the study through PCM referrals and posted advertisements. After a minimum of 6 hours post-vaginal delivery or 24 hours post caesarean section subjects will be given treatment according to their randomization group. Subjects will be assessed on pain control, overall satisfaction with pain management, and the amount of pharmacological pain medications used. Safety of measures will also be assessed to include infection rates, syncope, vertigo, and hypotension.

DETAILED DESCRIPTION:
Screening Visit:

* Obtain signed Informed Consent document and HIPAA Authorization.
* Review past medical history in Armed Forces Health Longitudinal Technology Application (AHLTA) to verify the inclusion/exclusion criteria and including previous encounter, vital signs review, medication list, co-morbidities, demographics, problems list, prior obstetric history, and note any prior acupuncture received.
* Record: Date of birth, age, gender, race, ethnicity, last 4 of social security number, current email address.

Randomization: Subjects will then be randomized into one of two groups by one of the Research Coordinators using a random number generator:

* Group 1: Standard of care only.
* Group 2: Standard of care plus Battlefield acupuncture at treatment sites Cingulate gyrus, thalamus, omega 2, shen-men, point zero in both ears (see figures 1-5). The 5 needles will remain in each ear for up to 7 days or allowed to fall out on their own (the patient will be instructed not to remove the needles).
* Subject's ears will be cleansed with an alcohol swab
* Subjects will be given a handout of standard BFA Discharge Instructions including what an infection looks like and what to do in the event of an infection (see attached).

Visit 1: Will occur after a minimum of 6 hours post vaginal birth (up until hospital discharge) to avoid disturbing maternal infant bonding or a minimum of 24 hours post caesarean section to avoid confounding with the anesthesia:

* Subject will be given treatment according to their randomization group.
* All subjects, regardless of randomization group, will be instructed to have no heavy meals, no excessive hot or cold foods, no heavy exercise or intercourse, and no alcohol for 6 hours.
* Satisfaction with post-partum pain management will be assessed with the following questions:
* On a scale of 0 to 10, how satisfied were you with your pain management after delivery? (dissatisfied 0 - 10 very satisfied)
* Would you use auricular acupuncture for future pain management? (Yes or no) (for those in the acupuncture group only)
* On a scale of 0-10, with 10 being the worst pain, what is your level of pain?

In hospital data collection: Data will be collected each day until the patient has been discharged from the hospital. Subjects will be contacted either in person or via phone and the hospital stay will vary from patient to patient:

* We will review the subject's medical record and record RN Recorded Pain assessments, Delivery method (either Caesarean section or spontaneous vaginal delivery), Delivery complications (vaginal lacerations, use of episiotomy, operative vaginal delivery, shoulder dystocia, post-partum hemorrhage), Birth weight, Maternal Parity, and record what pain medications they are taking.
* We will ask subjects if they prefer to be contacted in-person or via telephone while in the hospital.
* Satisfaction with post-partum pain management will be assessed with the following questions:
* On a scale of 0 to 10, how satisfied were you with your pain management after delivery? (dissatisfied 0 - 10 very satisfied)
* Would you use auricular acupuncture for future pain management? (Yes or no) (for those in the acupuncture group only)
* On a scale of 0-10, with 10 being the worst pain, what is your level of pain?
* Are the needles still in place? If yes, how many in each ear?

Post hospital discharge: Each day up until 10 days post Visit 1. Subjects will be contacted phone and the following information will be collected:

* Satisfaction with post-partum pain management will be assessed with the following questions:
* On a scale of 0 to 10, how satisfied were you with your pain management after delivery? (dissatisfied 0-10 very satisfied)
* Would you use auricular acupuncture for future pain management? (Yes or no) (for those in the acupuncture group only)
* On a scale of 0-10, with 10 being the worst pain, what is your level of pain? • We will record what pain medications they are taking including drug name, strength, and total doses since discharge from the hospital.

ELIGIBILITY:
THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY.

Inclusion:

* Post-partum female (DoD beneficiaries).
* Age 18 years or older
* Pain score rating post-delivery of greater or equal to 4/10.

Exclusion:

* Absence of one or more ears
* Active cellulitis of ear
* Ear anatomy precluding identification of acupuncture landmarks
* Non-English speaking
* Use of Hearing Aids that preclude the use of ear acupuncture
* Known allergy to gold

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2018-05-20 (Actual); Study Completion 2018-05-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Kim, MD, Principal Investigator — Mike O'Callaghan Federal Medical Center
Locations (1):
- Mike O'Callaghan Federal Medical Center, Nellis Air Force Base, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Deussen AR, Ashwood P, Martis R, Stewart F, Grzeskowiak LE. Relief of pain due to uterine cramping/involution after birth. Cochrane Database Syst Rev. 2020 Oct 20;10(10):CD004908. doi: 10.1002/14651858.CD004908.pub3. PMID 33078388
- [Derived] Zimpel SA, Torloni MR, Porfirio GJ, Flumignan RL, da Silva EM. Complementary and alternative therapies for post-caesarean pain. Cochrane Database Syst Rev. 2020 Sep 1;9(9):CD011216. doi: 10.1002/14651858.CD011216.pub2. PMID 32871021

RESULTS

PARTICIPANT FLOW:
Groups:
- Battlefield Auricular Acupuncture: Standard of Care plus Battlefield Auricular Acupuncture
  Battlefield Auricular Acupuncture
Period: Overall Study
Arm/Group | Standard of Care | Battlefield Auricular Acupuncture
Started | 33 | 37
Completed | 33 | 37
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard of Care | Battlefield Auricular Acupuncture | Total
Number analyzed (Participants) | 33 | 37 | 70
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 33 | 37 | 70
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 37 | 70
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 5 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 4 | 5
  White | 25 | 23 | 48
  More than one race | 6 | 4 | 10
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 33 | 37 | 70

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Achieved 50% Sustained Pain Reduction
Description: measured daily from days 0-11.
Time Frame: 12 days
Measure: Number; unit: # of subjects with 50% pain reduction
Arm/Group | Standard of Care | Battlefield Auricular Acupuncture
Number analyzed (Participants) | 33 | 37
# of subjects with 50% pain reduction
  day 0 | 0 | 0
  day 1 | 2 | 6
  day 2 | 3 | 9
  day 3 | 4 | 11
  day 4 | 8 | 12
  day 5 | 12 | 15
  day 6 | 16 | 17
  day 7 | 17 | 21
  day 8 | 20 | 22
  day 9 | 24 | 26
  day 10 | 25 | 26
  day 11 | 28 | 27

2. Secondary Outcome: Morphine Equivalent Use
Description: morphine equivalent units (total mg)
Time Frame: 12 days
Measure: Mean (Standard Deviation); unit: total mg
Arm/Group | Standard of Care | Battlefield Auricular Acupuncture
Number analyzed (Participants) | 33 | 37
total mg | 88 (58) | 82 (113)

ADVERSE EVENTS:
Time Frame: 12 days
Arm/Group | Standard of Care | Battlefield Auricular Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/37
Other Adverse Events (participants affected / at risk) | 0/33 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-29): https://cdn.clinicaltrials.gov/large-docs/86/NCT02526186/Prot_SAP_000.pdf